CLINICAL TRIAL: NCT02821689
Title: Randomized Controlled Trial of Pirfenidone in Patients With Progressive Interstitial Lung Disease Associated With Clinically Amyopathic Dermatomyositis
Brief Title: Pirfenidone in Progressive Interstitial Lung Disease Associated With Clinically Amyopathic Dermatomyositis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Shuang Ye, Executive Director, Dept. Rheumatology, Renji Hospital South Campus, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RenJi-ADM
Record Dates: First submitted 2016-06-21; First posted 2016-07-01 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Dermatopolymyositis; Interstitial Lung Disease
Keywords: Dermatopolymyositis; Interstitial lung disease; Pirfenidone
MeSH Terms: conditions — Dermatomyositis; Lung Diseases, Interstitial | interventions — pirfenidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pirfenidone (Experimental): Eligible participants for clinical trial were randomized in a 2:1 ratio to pirfenidone/blank add-on. Pirfenidone was administered in three divided doses (200mg tid), and increased to the manufacturer's instructed target dose (600mg tid) over a 2-week period. Investigators were allowed to adjust the dose according to the participants' tolerance.
  Interventions: Drug: Pirfenidone
- Blank (No Intervention): Eligible participants for clinical trial were randomized in a 2:1 ratio to pirfenidone/blank add-on.

INTERVENTIONS:
Drug: Pirfenidone — Pirfenidone was administered in three divided doses (200mg tid), and increased to the manufacturer's instructed target dose (600mg tid) over a 2-week period. The maximum dose was maintained throughout the study in patients who tolerated it.
  Arms: pirfenidone

SUMMARY:
Interstitial lung disease (ILD) is a common complication of dermatomyositis (DM) with prevalence up to 65%, and is considered to be one of the determining factors of prognosis. Clinical amyopathic dermatomyositis (CADM), which is a special phenotype of DM, with characteristic cutaneous manifestations but no or only subclinical myopathy. Many studies, mainly from Asia, including ours, have demonstrated that these patients with CADM tend to develop a rapidly progressive ILD (RPILD) and have a poor response to conventional therapy, such as high-dose corticosteroids and immunosuppressants, leading to lethal outcome with a 6-month survival rate of less than 50%.

Pirfenidone, a new oral antifibrotic agent, has been approved for the treatment of idiopathic pulmonary fibrosis (IPF). Randomized controlled trials of pirfenidone in patients with IPF suggested that it could ameliorate pulmonary function decline and improve the progression-free survival. Its utility in connective tissue disease (CTD) related ILD has been implicated, but no evidence has yet demonstrated its efficacy. Therefore, the investigators conduct this study to evaluate the possible therapeutic effects of pirfenidone on RPILD associated with CADM.

ELIGIBILITY:
Inclusion Criteria:

* Willingness of the subject to participate in the study, proven by signing the informed consent;
* All participants fulfilled the provisional diagnosis of CADM according to the modified Sontheimer's criteria.
* The course of ILD is longer than 3 months, but shorter than 6 months, presenting as increase in level of dyspnea, and worsening of fibrosis on pulmonary HRCT with >10% increase of HRCT score, and/or decrease in %FVC by >10% absolute value.

Exclusion Criteria:

* Participants who are unwilling to sign the inform consent;
* The course of participants ever treated with biologics including basiliximab, or malignancy-associated CADM or overlapped with other CTD, or with alanine transaminase more than 2 times the upper normal limits;
* Pregnancy or lactation.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
changes of 12-month survival from the onset of ILD | 12 months
  the effect of pirfenidone on improving the survival rate

SECONDARY OUTCOMES:
changes of high-resolution computed tomography (HRCT) scores from baseline at each visit | one year
  the influence of pirfenidone on pulmonary interstitial changes
changes of pulmonary function test from baseline at each visit | one year
  the influence of pirfenidone on pulmonary function changes

CONTACTS AND LOCATIONS:
Overall Officials: Shuang Ye, MD, Principal Investigator — RenJi Hospital
Locations (1):
- Department of Rheumatology, Ren Ji Hospital South Campus, School of Medicine, Shanghai JiaoTong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided